CLINICAL TRIAL: NCT02711150
Title: Efficacy of the Epidural Positioning Device (EPD) on Optimising the Acoustic Target Window for Neuraxial Needle Placement
Brief Title: Effect of EPD on the Lumbar Acoustic Window at Term Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: 107422
Record Dates: First submitted 2016-01-26; First posted 2016-03-17 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Effects of; Anesthesia, Spinal and Epidural, in Pregnancy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPD Measurements (Experimental): Intervention:
  PLL Length Measured through US will be done with the subject placed on the Epidural Positioning Device.
  Interventions: Device: PLL Length Measured through US
- Flexed Position Measurements (Active Comparator): Intervention:
  PLL Length Measured through US will be done with the subject placed in a "flexed" lumbar spine position.
  Interventions: Device: PLL Length Measured through US

INTERVENTIONS:
Device: PLL Length Measured through US — The PLL will be measured for each allocated position: EPD or Flexed Position
  Other Names: PLL length

SUMMARY:
The purpose of this study is to assess whether application of an epidural positioning device to a parturient seated for neuraxial anaesthesia increase the size of the paramedian target area for neuraxial needle insertion. Lumbar ultrasonography will be performed in 30 pregnant women in two seated positions: (P1), lumbar flexion; and (P2), as in P1 with the epidural positioning device applied. For each position, the size of the 'target area', defined as the visible length of the posterior longitudinal ligament will be measured at the L3-L4 interspace.

DETAILED DESCRIPTION:
Thirty term pregnant women will be recruited. Signed informed consent will be obtained from all subjects and demographic details, including age, weight, height and body mass index (BMI) will be documented. Randomization and blinding: Randomization will not be performed in this study, because each patient is their own control Interventions: Two experienced operators who have previously performed several hundred landmark-guided and ultrasound-assisted neuraxial blocks will perform the clinical and ultrasound examination.. The patient will then be placed in each of the positions described below. While in each of the positions an ultrasound (US) probe will be placed at level L3- L4 at the paramedian position to visualize the paravertebral longitudinal ligament (PLL) . These measurements will be recorded by an observer. In both phases (first US operator and second US operator ), 2 ultrasound measurements will be made for each of the following positions at 1 lumbar level in the paramedian view. These measurements will be made with the patient in the following positions: • Sitting position, feet supported with back flexed. • Sitting position, feet supported and arms supported through the application of an epidural positioning device. All images will be assigned a number based on a random number generator to remove any identifying data, including volunteer number, date, time, and position. The PLL will be remeasured on every saved image by two separate anesthesiologists ('readers') who are not involved with any previous data collection but are members of the study team. Both will be blinded to the number allocation and each other's measured values. This aim to remove any bias by the 'scanning' anesthesiologists and test for reproducibility in the measurement of the PLL, between 'readers'. A statistician calculated a minimum sample size of 30 subjects, in order to demonstrate significant change in the mean length of the PLL (acoustic target area), in any of the two positions. This estimation was based on data derived from a similar study, which had used a minimum sample size of 16 subjects, with a 1 mm mean change in 'needle target area' dimensions, a 1 mm standard deviation (SD), and an alpha of 0.05 with a power of 90 % [1, 2].

ELIGIBILITY:
Inclusion Criteria:

* Female Patients
* Term Pregnancy (>37 weeks)
* 18 years or older
* Non-labouring patients, admitted for a cesarean delivery

Exclusion Criteria:

* Allergy to ultrasound jelly
* Spinal Deformities
* Active Labour
* Presence of Epidural Catheter for Labour Analgesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2016-10-07 (Actual)

PRIMARY OUTCOMES:
Increase in PLL with the application of an EPD | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Indu Singh, MD, FRCPC, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones AR, Carle C, Columb M. Effect of table tilt on ligamentum flavum length measured using ultrasonography in pregnant women*. Anaesthesia. 2013 Jan;68(1):27-30. doi: 10.1111/anae.12006. Epub 2012 Oct 22. PMID 23088766
- [Background] Grau T, Leipold RW, Horter J, Conradi R, Martin EO, Motsch J. Paramedian access to the epidural space: the optimum window for ultrasound imaging. J Clin Anesth. 2001 May;13(3):213-7. doi: 10.1016/s0952-8180(01)00245-8. PMID 11377160